CLINICAL TRIAL: NCT05621655
Title: A Phase II Randomized, Double-blind, Placebo-controlled Clinical Trial to Evaluate the Safety and Immunogenicity of Recombinant Trivalent Subunit Rotavirus Vaccine in Healthy Infants Aged 6-12 Weeks and Healthy Toddlers Aged 7-71 Months
Brief Title: Safety and Immunogenicity Study of Recombinant Trivalent Rotavirus Subunit Vaccine in Healthy Infants and Toddlers
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: MAXVAX Biotechnology Limited Liability Company (Industry)
Collaborators: Henan Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MKKCT2021002
Record Dates: First submitted 2022-11-07; First posted 2022-11-18 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Rotavirus Infections; Rotavirus Gastroenteritis
Keywords: Rotavirus; Gastroenteritis
MeSH Terms: conditions — Rotavirus Infections; Gastroenteritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (12):
- Mid dose in toddlers (7-71 months old, 3 doses) (Experimental): Mid dose recombinant trivalent rotavirus subunit vaccine in toddlers aged 7-71 months on Day 0, 28 and 56, intramuscularly injected.
  Interventions: Biological: Mid dose Recombinant Trivalent Subunit Rotavirus Vaccine
- Mid dose in toddlers (7-71 months old, 2 doses) (Experimental): Mid dose recombinant trivalent rotavirus subunit vaccine in toddlers aged 7-71 months on Day 0 and 28, intramuscularly injected.
  Interventions: Biological: Mid dose Recombinant Trivalent Subunit Rotavirus Vaccine
- High dose in toddlers (7-71 months old, 3 doses) (Experimental): High dose recombinant trivalent rotavirus subunit vaccine in toddlers aged 7-71 months on Day 0, 28 and 56, intramuscularly injected.
  Interventions: Biological: High dose Recombinant Trivalent Subunit Rotavirus Vaccine
- High dose in toddlers (7-71 months old, 2 doses) (Experimental): High dose recombinant trivalent rotavirus subunit vaccine in toddlers aged 7-71 months on Day 0 and 28, intramuscularly injected.
  Interventions: Biological: High dose Recombinant Trivalent Subunit Rotavirus Vaccine
- Placebo in toddlers (7-71 months old, 3 doses) (Placebo Comparator): Placebo in toddlers aged 7-71 months on Day 0, 28 and 56, intramuscularly injected.
  Interventions: Biological: Placebo
- Placebo in toddlers (7-71 months old, 2 doses) (Placebo Comparator): Placebo in toddlers aged 7-71 months on Day 0 and 28, intramuscularly injected.
  Interventions: Biological: Placebo
- Mid dose in infants (6-12 weeks of age, 3 doses at 4-week intervals) (Experimental): Mid dose recombinant trivalent rotavirus subunit vaccine in infants aged 6-12 weeks on Day 0, 28 and 56, intramuscularly injected.
  Interventions: Biological: Mid dose Recombinant Trivalent Subunit Rotavirus Vaccine
- Mid dose in infants (6-12 weeks of age, 3 doses at 8-week intervals) (Experimental): Mid dose recombinant trivalent rotavirus subunit vaccine in infants aged 6-12 weeks on Day 0, 56 and 112, intramuscularly injected.
  Interventions: Biological: Mid dose Recombinant Trivalent Subunit Rotavirus Vaccine
- High dose in infants (6-12 weeks of age, 3 doses at 4-week intervals) (Experimental): High dose recombinant trivalent rotavirus subunit vaccine in infants aged 6-12 weeks on Day 0, 28 and 56, intramuscularly injected.
  Interventions: Biological: High dose Recombinant Trivalent Subunit Rotavirus Vaccine
- High dose in infants (6-12 weeks of age, 3 doses at 8-week intervals) (Experimental): High dose recombinant trivalent rotavirus subunit vaccine in infants aged 6-12 weeks on Day 0, 56 and 112, intramuscularly injected.
  Interventions: Biological: High dose Recombinant Trivalent Subunit Rotavirus Vaccine
- Placebo in infants (6-12 weeks of age, 3 doses at 4-week intervals) (Placebo Comparator): Placebo in infants aged 6-12 weeks on Day 0, 28 and 56, intramuscularly injected.
  Interventions: Biological: Placebo
- Placebo in infants (6-12 weeks of age, 3 doses at 8-week intervals) (Placebo Comparator): Placebo in infants aged 6-12 weeks on Day 0, 56 and 112, intramuscularly injected.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Mid dose Recombinant Trivalent Subunit Rotavirus Vaccine — 0.5 mL of vaccine containing a total of 60 µg of protein (20 µg of each P type) adjuvanted with 0.5 mg aluminum hydroxide.
  Arms: Mid dose in infants (6-12 weeks of age, 3 doses at 4-week intervals); Mid dose in infants (6-12 weeks of age, 3 doses at 8-week intervals); Mid dose in toddlers (7-71 months old, 2 doses); Mid dose in toddlers (7-71 months old, 3 doses)
Biological: High dose Recombinant Trivalent Subunit Rotavirus Vaccine — 0.5 mL of vaccine containing a total of 90 µg of protein (30 µg of each P type) adjuvanted with 0.5 mg aluminum hydroxide.
  Arms: High dose in infants (6-12 weeks of age, 3 doses at 4-week intervals); High dose in infants (6-12 weeks of age, 3 doses at 8-week intervals); High dose in toddlers (7-71 months old, 2 doses); High dose in toddlers (7-71 months old, 3 doses)
Biological: Placebo — 0.5 mL per dose, containing 0.5 mg aluminium hydroxide adjuvant.
  Arms: Placebo in infants (6-12 weeks of age, 3 doses at 4-week intervals); Placebo in infants (6-12 weeks of age, 3 doses at 8-week intervals); Placebo in toddlers (7-71 months old, 2 doses); Placebo in toddlers (7-71 months old, 3 doses)

SUMMARY:
The purpose of this study is to assess the immunogenicity, safety and immune persistence of recombinant trivalent rotavirus subunit vaccine in healthy infants aged 6-12 weeks and healthy toddlers aged 7-71 months.

DETAILED DESCRIPTION:
This clinical trial is aimed to evaluate the immunogenicity, safety and immune persistence of recombinant trivalent rotavirus subunit vaccine in Chinese healthy infants aged 6-12 weeks and healthy toddlers aged 7-71 months.The subjects will be divided into 12 subgroups. Two different immune regimens and two dose levels will be evaluated in each age group. Toddlers aged 7-71 months will receive two intramuscular injections on Day 0 and 28 or three intramuscular injections on Day 0, 28 and 56. Infants aged 6-12 weeks will receive three intramuscular injections on Day 0, 28 and 56 or Day 0, 56 and 112. Two dose (mid dose and high dose) will be included in each age group. To maintain blindness in the trial, in each age group with fixed immune regimen, subjects will be randomized in a 1:1:1 ratio to receive mid dose vaccine, high dose vaccine, or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy infants aged 6-12 weeks and healthy toddlers aged 7-71 months;
2. Legally acceptable representative (guardian) properly informed about the study and having signed the informed consent form (ICF).

Exclusion Criteria:

First dose exclusion criteria:

1. Axillary temperature >37.0℃ before vaccination;
2. Recepit of any rotavirus vaccine in the past;
3. History of intussusception or suffering from intussusception or history of any chronic gastrointestinal disease, including congenital malformations of the gastrointestinal tract that are likely to cause intussusception (such as Meckel's diverticulum);
4. Congenital malformations, developmental disorders, genetic defect, severe malnutrition, etc.;
5. Subjects aged 2 years or younger with history of dystocia, suffocation rescue, or nervous system damage;
6. Subjects aged 2 years or younger with history of premature birth (<37 weeks' gestation) or low birth weight (weight at birth of<2500 g);
7. History of convulsions, epilepsy and cerebral palsy, or mental illness and family history;
8. History of severe anaphylactic reaction to vaccination, or allergy to any components of the study vaccine;
9. Acute diseases (such as fever>39.0℃) or acute exacerbation of chronic disease within 3 days before vaccination;
10. Receipt of immune enhancement (including oral or intravenous immunoglobulin, but hepatitis B immunoglobulin is acceptable) or immunosuppressive therapy (continuous oral or intravenous infusion for more than 14 days) within 3 months;
11. Recepit of live attenuated vaccines within 14 days, or other vaccines within 7 days;
12. Congenital or acquired immunodeficiency, HIV infection, lymphoma, leukemia, systemic lupus erythematosus (SLE), juvenile rheumatoid arthritis (JRA), or other autoimmune diseases;
13. History of coagulation abnormalities (such as lack of blood coagulation factors, blood coagulopathy);
14. Primary and secondary impairment of immune function (history of thyroid, pancreas, liver, spleen resection, or treatment due to thyroid disease within the past 12 months);
15. Concurrent participation or plan to participate in another clinical trial throughout the study;
16. According to the judgment of the investigator, the subject has any other factors that are not suitable for participating in the clinical trial.

    Subsequent vaccination exclusion criteria:
17. Severe allergic reaction after the previous injection of study vaccine;
18. Serious adverse reactions that are causally related to the previous vaccination;
19. After the first vaccination, subjects with newly discovered or newly happened diseases that meet the first dose exclusion criteria will be determined by the investigator whether to continue participating the study;
20. Other reasons for exclusion judged by the investigator.

Ages: 6 Weeks to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1512 (Actual)
Dates: Start 2023-01-08 (Actual); Primary Completion 2023-04-29 (Actual); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
The incidence of adverse events | Within 30 minutes after each vaccination
  Incidence of adverse events within 30 minutes after each dose. The severity of solicited and unsolicited adverse events will be graded from grade 1 to grade 4, other adverse events will be graded from grade 1 to grade 5.
The incidence of adverse events | Within 14 days after each vaccination
  Incidence of adverse events within 14 days after each dose. The severity of solicited and unsolicited adverse events will be graded from grade 1 to grade 4, other adverse events will be graded from grade 1 to grade 5.
The incidence of adverse events | Day 15 to 28/30 after each vaccination
  Incidence of adverse events Day 15 to 28/30 after each dose. The severity of solicited and unsolicited adverse events will be graded from grade 1 to grade 4, other adverse events will be graded from grade 1 to grade 5.
The incidence of adverse events | Within 28/30 days after each vaccination
  Incidence of adverse events within 28/30 days after each dose. The severity of solicited and unsolicited adverse events will be graded from grade 1 to grade 4, other adverse events will be graded from grade 1 to grade 5.
Geometric Mean Titers (GMT) of anti-P[4], anti-P[6], anti-P[8] rotavirus Immunoglobulin A (IgA) | Day 30 after the last vaccination
  Measured by ELISA at baseline and 30 days after the last vaccination.
Geometric Mean Titers (GMT) of anti-P[4], anti-P[6], anti-P[8] rotavirus Immunoglobulin G (IgG) | Day 30 after the last vaccination
  Measured by ELISA at baseline and 30 days after the last vaccination.
Geometric Mean Titers (GMT) of anti-P[4], anti-P[6], anti-P[8] rotavirus neutralizing antibody | Day 30 after the last vaccination
  Neutralizing antibodies will be measured by Micro serum neutralization test at baseline and 30 days after the last vaccination.
Seroconversion rates of anti-P[4], anti-P[6], anti-P[8] rotavirus IgA | Day 30 after the last vaccination
  Seroconversion is defined as a ≥ 4-fold rise in IgA titer compared with Baseline.
Seroconversion rates of anti-P[4], anti-P[6], anti-P[8] rotavirus IgG | Day 30 after the last vaccination
  Seroconversion is defined as a ≥ 4-fold rise in IgG titer compared with Baseline.
Seroconversion rates of anti-P[4], anti-P[6], anti-P[8] rotavirus neutralizing antibody | Day 30 after the last vaccination
  Seroconversion is defined as a ≥ 2.7-fold rise in neutralizing antibody titer compared with Baseline.

SECONDARY OUTCOMES:
Incidence of serious adverse events (SAE) | From the first vaccination to 12 months after the last vaccination.
  Incidence of serious adverse events throughout the study.
Geometric Mean Titers (GMT) of anti-P[4], anti-P[6], anti-P[8] rotavirus IgA | Day 90 after the last vaccination
  Measured by ELISA.
Geometric Mean Titers (GMT) of anti-P[4], anti-P[6], anti-P[8] rotavirus IgA | Day 180 after the last vaccination
  Measured by ELISA.
Geometric Mean Titers (GMT) of anti-P[4], anti-P[6], anti-P[8] rotavirus IgA | Day 360 after the last vaccination
  Measured by ELISA.
Geometric Mean Titers (GMT) of anti-P[4], anti-P[6], anti-P[8] rotavirus IgG | Day 90 after the last vaccination
  Measured by ELISA.
Geometric Mean Titers (GMT) of anti-P[4], anti-P[6], anti-P[8] rotavirus IgG | Day 180 after the last vaccination
  Measured by ELISA.
Geometric Mean Titers (GMT) of anti-P[4], anti-P[6], anti-P[8] rotavirus IgG | Day 360 after the last vaccination
  Measured by ELISA.
Geometric Mean Titers (GMT) of anti-P[4], anti-P[6], anti-P[8] rotavirus neutralizing antibody | Day 90 after the last vaccination
  Neutralizing antibodies will be measured by Micro serum neutralization test.
Geometric Mean Titers (GMT) of anti-P[4], anti-P[6], anti-P[8] rotavirus neutralizing antibody | Day 180 after the last vaccination
  Neutralizing antibodies will be measured by Micro serum neutralization test.
Geometric Mean Titers (GMT) of anti-P[4], anti-P[6], anti-P[8] rotavirus neutralizing antibody | Day 360 after the last vaccination
  Neutralizing antibodies will be measured by Micro serum neutralization test.
Seroconversion rates of anti-P[4], anti-P[6], anti-P[8] rotavirus IgA | Day 90 after the last vaccination
  Seroconversion is defined as a ≥ 4-fold rise in IgA titer compared with Baseline.
Seroconversion rates of anti-P[4], anti-P[6], anti-P[8] rotavirus IgA | Day 180 after the last vaccination
  Seroconversion is defined as a ≥ 4-fold rise in IgA titer compared with Baseline.
Seroconversion rates of anti-P[4], anti-P[6], anti-P[8] rotavirus IgA | Day 360 after the last vaccination
  Seroconversion is defined as a ≥ 4-fold rise in IgA titer compared with Baseline.
Seroconversion rates of anti-P[4], anti-P[6], anti-P[8] rotavirus IgG | Day 90 after the last vaccination
  Seroconversion is defined as a ≥ 4-fold rise in IgG titer compared with Baseline.
Seroconversion rates of anti-P[4], anti-P[6], anti-P[8] rotavirus IgG | Day 180 after the last vaccination
  Seroconversion is defined as a ≥ 4-fold rise in IgG titer compared with Baseline.
Seroconversion rates of anti-P[4], anti-P[6], anti-P[8] rotavirus IgG | Day 360 after the last vaccination
  Seroconversion is defined as a ≥ 4-fold rise in IgG titer compared with Baseline.
Seroconversion rates of anti-P[4], anti-P[6], anti-P[8] rotavirus neutralizing antibody | Day 90 after the last vaccination
  Seroconversion is defined as a ≥ 2.7-fold rise in neutralizing antibody titer compared with Baseline.
Seroconversion rates of anti-P[4], anti-P[6], anti-P[8] rotavirus neutralizing antibody | Day 180 after the last vaccination
  Seroconversion is defined as a ≥ 2.7-fold rise in neutralizing antibody titer compared with Baseline.
Seroconversion rates of anti-P[4], anti-P[6], anti-P[8] rotavirus neutralizing antibody | Day 360 after the last vaccination
  Seroconversion is defined as a ≥ 2.7-fold rise in neutralizing antibody titer compared with Baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Yanxia Wang, Principal Investigator — Henan Center for Disease Control and Prevention
Locations (2):
- China (2):
  - Shangqiu Liangyuan District Center for Disease Control and Prevention, Shangqiu, Henan
  - Ningling County Center for Disease Control and Prevention, Shangqiu, Henan

IPD SHARING:
Plan to Share IPD: No